CLINICAL TRIAL: NCT05734482
Title: Phase I Comparison of Pharmacokinetics, Safety, and Immunogenicity of CMAB015 Injection and Cosentyx in a Randomized, Double-blind, Parallel Controlled, Single-dose Study in Healthy Chinese Male Subjects
Brief Title: Pharmacokinetic, Safety and Immunogenicity Study of CMAB015 and Cosentyx in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMAB015-001
Record Dates: First submitted 2023-01-29; First posted 2023-02-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Biological: CMAB015 Biological: Cosentyx（Secukinumab ）
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biosimilar Product (Experimental): CMAB015 150 mg Subcutaneous injection in upper arm
  Interventions: Biological: Secukinumab
- Reference Product (Active Comparator): Cosentyx（Secukinumab ） 150 mg Subcutaneous injection in upper arm
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: Secukinumab — for subcutaneous injection only

SUMMARY:
This is a randomized, double-blinded, controlled Phase I study of CMAB015 administered by subcutaneous injection. This study will characterize the pharmacokinetic, safety and immunogenicity of CMAB015 versus Cosentyx（Secukinumab ） in healthy male subjects after a single dose.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-controlled, single-dose phase I clinical study in healthy Chinese male subjects. A total of 130 subjects were planned to be enrolled and randomly assigned to the test group or the control group in a 1:1 ratio. Subjects in both groups received a single upper arm subcutaneous injection of CMAB015 or Cosentyx（Secukinumab） 150 mg, respectively. Subjects in both groups were observed for 112 days after administration to evaluate similarities in pharmacokinetics, safety, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age ranged 18 to 45 years (both inclusive)；
2. Subjects with body weight of ≥50 kg and ≤ 75 kg and BMI ≥18 and <28 kg/m2 ;
3. Subjects and their partners were willing to use medically approved contraceptive methods within 6 months of study administration, partners did not plan to become pregnant, subjects did not plan to donate sperm；
4. The subjects have the ability to understand the full characteristics and objectives of the study, including the possible risks and side effects of the study; Moreover, the subjects can communicate well with researchers and complete the research according to the regulations；
5. Subjects voluntarily sign ICF prior to the study.

Exclusion Criteria:

1. After comprehensive examination (vital signs, physical examination, electrocardiogram, chest radiography, abdominal B-ultrasound, blood routine, urine routine, blood biochemistry, etc.), any examination item was judged abnormal by the investigator and had clinical significance;
2. Patients with serious diseases such as cardiovascular system, endocrine system, nervous system, digestive system, respiratory system, genitourinary system, hematopoietic system, immune system, or any of the above diseases；
3. Patients with currently active infected diseases；
4. Subjects with past or current inflammatory bowel disease;
5. History of malignant neoplasms within the last 5 years (other than completely resected basal cell or squamous cell carcinoma of the skin in situ)；
6. Any one of HBV surface antigen, HCV antibody, HIV antibody, treponema pallidum antibody positive；
7. Subjects with T-SPOT test positive；
8. Those who smoked more than 5 cigarettes per day in the 6 months before screening and did not cooperate with smoking bans during the study period；
9. Alcoholics，or participants who consumed more than 14 units of alcohol per week (1 unit = 17.7mL ethanol, i.e., 1 unit = 357mL 5% beer or 43mL 40% liquor or 147mL 12% wine) during the preceding 3 months were screened，or who have positive result in blood-test of alcohol or not willing to ban alcohol；
10. Drug abusers, or drug users in the 3 months prior to screening, or excessive daily consumption of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250mL) in the 3 months prior to screening, or positive urine drug screening；
11. Surgery within 4 weeks prior to screening; Or plan to have surgery during the study period；
12. Use of any prescription drug, over-the-counter drug or health product within 4 weeks prior to screening, or prior use of such drug or health product within 5 half-lives, whichever is longer；
13. Those who have used any biological agent, including live vaccine, in the 3 months prior to screening, or who plan to receive live vaccine during the study period；
14. Anti-il-17 antibody active ingredient, excipients or latex allergy；
15. Those with anti-IL-17 antibody and anti-drug antibody positive；
16. Those who have been enrolled in other clinical studies or less than 3 months since the end of the most recent clinical study；
17. Those who had lost blood or donated at least 400 mL in the 3 months prior to the trial, or had lost blood or donated at least 200 mL in the 1 month prior to screening, or planned to donate blood during the trial；
18. Those who Can not tolerate venipunction, has a history of dizziness of needle and blood；
19. Those who have special dietary requirements, or can not accept uniform diet；
20. Other conditions considered inappropriate to be included in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Zero (0) Hours Extrapolated to infinite time | up to 2688 hours
  Area Under the Plasma Concentration-time Curve From Zero (0) Hours Extrapolated to infinite time After the Single injection of CMAB015/Cosentyx
Maximum Concentration of Secukinumab | up to 2688 hours
  Maximum Concentration of Secukinumab After the Single Injection of CMAB015/Cosentyx

SECONDARY OUTCOMES:
Time to Maximum Concentration of Secukinumab | up to 2688 hours
  Time to Maximum Concentration of Secukinumab after the Single Injection of CMAB015/Cosentyx
Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 2688 Hours | up to 2688 hours
  Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 2688 Hours After the Single Injection of CMAB015/Cosentyx
Half time | up to 2688 hours
  Half-time after the Single Injection of CMAB015/Cosentyx
Clearance Rate | up to 2688 hours
  Clearance Rate after the Single Injection of CMAB015/Cosentyx
Apparent Volume of Distribution | up to 2688 hours
  Apparent Volume of Distribution after the Single Injection of CMAB015/Cosentyx
Terminal phase elimination rate constant | up to 2688 hours
  Terminal phase elimination rate constant after the Single Injection of CMAB015/Cosentyx
anti-drug antibodies(ADA) | up to 2688 hours
  ADA Positive Rate after the Single Injection of CMAB015/Cosentyx
Neutralization antibodies(Nab) | up to 2688 hours
  Neutralizing Antibody Positive Rate after the Single Injection of CMAB015/Cosentyx
Percentage of participants with Adverse Events | up to 2688 hours
  Total Frequency of Adverse Events/Serious Adverse Events Within the Whole Time of the Study

CONTACTS AND LOCATIONS:
Overall Officials: Hu Wei, Doctor, Principal Investigator — The Second Hospital of Anhui University
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yao F, Wang C, Ding J, Zhang Q, Zheng L, Zhang Q, Yang T, Zhang X, Shan Y, Hou S, Wang H, Zhou R, Hu W. A Randomized, Double-Blind, Parallel-Group Phase I Study Comparing the Pharmacokinetics, Safety, and Immunogenicity of CMAB015, a Candidate Secukinumab Biosimilar, with Its Reference Product Cosentyx(R) in Healthy Chinese Male Subjects. Drug Des Devel Ther. 2024 Aug 29;18:3891-3901. doi: 10.2147/DDDT.S470619. eCollection 2024. PMID 39224901